CLINICAL TRIAL: NCT00940381
Title: A Phase I Trial of Sirolimus and Cetuximab in Patients With Advanced Malignancies
Brief Title: Sirolimus and Cetuximab in Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0226; NCI-2012-01271 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-07-14; First posted 2009-07-16 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2014-05

CONDITIONS: Advanced Cancer
Keywords: Advanced Malignancies; Sirolimus; Rapamune; Cetuximab; C225; Erbitux; IMC-225
MeSH Terms: interventions — Sirolimus; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sirolimus + Cetuximab (Experimental): Sirolimus beginning dose 3 mg by mouth on Day 1, and 1 mg on Days 2 - 28 for a 28 day cycle. Cetuximab Beginning dose 100 mg/m^2 by vein over two hours on Day 1, and 65 mg/m^2 on Days 8, 15 and 22 for a 28 day cycle.
  Interventions: Drug: Sirolimus; Drug: Cetuximab

INTERVENTIONS:
Drug: Sirolimus — Beginning dose 3 mg by mouth on Day 1, and 1 mg on Days 2 - 28 for a 28 day cycle.
  Other Names: Rapamune
Drug: Cetuximab — Beginning dose 100 mg/m^2 by vein over two hours on Day 1, and 65 mg/m^2 on Days 8, 15 and 22 for a 28 day cycle.
  Other Names: C225; Erbitux; IMC-225

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of the combination of sirolimus and cetuximab that can be given to patients with advanced cancer. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Cetuximab is designed to prevent or slow down the growth of cancer cells by blocking protein on the surface of the cancer cell, called the epidermal growth factor receptor (EGFR).

Sirolimus is designed to block a protein called mTOR inside the cancer cell. This may interfere with the growth or spread of cancer cells or possibly kill the cancer cells.

Study Drug Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of cetuximab and sirolimus based on when you joined this study. Up to 9 dose levels of cetuximab and sirolimus will be tested. Three (3) to 9 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of the combination of cetuximab and sirolimus is found.

Once the highest tolerated dose of the combination of cetuximab and sirolimus is found, 2 groups of additional participants (Group 1 and Group 2, each of 14 participants) will be enrolled and receive the study drugs at that dose level. Another 14 participants with the non-small lung and head and neck cancer will receive the study drug at that dose level, as well.

Study Drug Administration:

Each study "cycle" is 28 days.

Everyday, you will take sirolimus by mouth 1 time a day. You should take it at about the same time each day with food and a cup of water.

On Days 1, 8, 15, and 22 of each cycle, you will receive cetuximab by vein over 2 hours. If the first dose is well tolerated, you will receive the next dose over 1 hour.

Study Visits:

At every study visit, you will be asked about any current health conditions you have, drugs you are taking, and if you have experienced any side effects.

Between Days 8 and 15 of Cycle 1, the following tests and procedures will be performed:

-If you are enrolled in a Group 2 of the highest drug combination dose, you will have a tumor biopsy and your blood (about 1-3 tablespoons) will be drawn for pharmacodynamic (PD) testing.

About Days 8 and 22 of Cycle 1, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests.

About Day 15 of Cycle 1, blood (about 2 teaspoons) will be drawn for routine tests.

About Day 22 of Cycles 2 and then every 1-2 cycles, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests.

Every 4 weeks, you will have a blood (about 1 teaspoon) drawn or urine collected for pregnancy test if you are able to become pregnant.

Every 8 weeks, you will have an x-ray, CT scan, MRI, and/or PET/CT to check the status of the disease. The study doctor thinks it is needed, they will be performed more often.

Length of Study:

You may stay on study for as long as you are benefitting. You will be taken off study if you experience intolerable side effects, the study doctor thinks it is in your best interest, or the cancer gets worse.

End-of-Study Visit:

About 28 days after the last dose of study drugs, you will have an end-of-study visit. At this visit, the following tests or procedures may be performed:

* You will have a physical exam, including measurement of your vital signs.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* If the doctor thinks it is needed, you will have an x-ray, CT, MRI, and/or PET/CT to check the status of the disease.

This is an investigational study. Sirolimus is FDA approved and commercially available as an anti-rejection drug for kidney transplant recipients. Cetuximab is FDA approved and commercially available for the treatment of colorectal and head/neck cancers. The combination of these drugs is investigational.

Up to 137 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced or metastatic cancer that is refractory to standard therapy, relapsed after standard therapy, or who have no standard therapy available that improves survival by at least three months.
2. Patients must be >/= 3 weeks beyond treatment with a cytotoxic chemotherapy regimen, or therapeutic radiation, or major surgery. Patients may have received palliative localized radiation immediately before or during treatment providing radiation is not delivered to the only site of disease being treated under this protocol. For biologic/targeted agents patients must be >/= 5 half-lives or >/= 3 weeks form the last dose (whichever comes first).
3. Eastern Cooperative Oncology Group (ECOG) performance status </= 3.
4. Patients must have normal organ and marrow function defined as: absolute neutrophil count >/= 1,000/mL; platelets >/=50,000/mL; creatinine </= 3 X upper limit of normal (ULN); total bilirubin </= 2.0; ALT(SGPT) </= 5 X ULN; Exception for patients with liver metastasis: total bilirubin </= 3 x ULN; ALT(SGPT) </= 8 X ULN; cholesterol </= 350 mg/dL; triglycerides </= 400 mg/dL.
5. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 30 days after the last dose.
6. Patients with colorectal cancer with Kirsten rat sarcoma (kRAS) mutations (mutational status must be available prior to entering the study)
7. Patients must be able to understand and be willing to sign a written informed consent document.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, uncontrolled asthma, need for hemodialysis, need for ventilatory support.
2. Pregnant or lactating women.
3. History of hypersensitivity to cetuximab, murine products, or any component of the formulation.
4. History of hypersensitivity to sirolimus.
5. History of hypersensitivity to any component of the formulation.
6. Patients with colorectal cancer with kRAS mutations. (mutational status must be available prior to entering the study)
7. Patients unwilling or unable to sign informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2009-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Dose-Limiting Toxicities (DLT) of Combination Treatment with Sirolimus and Cetuximab | 4 weeks
  MTD defined by DLTs that occur in the first cycle (4 weeks). DLT defined as any clinically grade 3 or 4 non-hematologic toxicity as defined in the NCI CTC v3.0, expected and believed to be related to the study medications (except nausea and vomiting, electrolyte imbalances responsive to appropriate regimens or alopecia), any grade 4 hematologic toxicity lasting at least 3 weeks or longer (as defined by the NCI-CTC v3.0) or associated with bleeding and/or sepsis; any grade 4 nausea or vomiting > 5 days despite maximum anti-nausea regimens, and any other grade 3 non-hematologic toxicity including symptoms/signs of vascular leak or cytokine release syndrome; or any severe or life-threatening complication or abnormality not defined in the NCI-Common Toxicity Criteria for Adverse Effects (CTCAE) v3.0 that is attributable to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Filip Janku, MD,PHD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org